CLINICAL TRIAL: NCT04612127
Title: Nutritional Clinical Trial to Evaluate the Efficacy of Daily Consumption for 12 Weeks of a Spinach Extract on Muscle Function in Subjects Over 50 Years of Age
Brief Title: Efficacy of the Consumption of a Spinach Extract on Muscle Function in Subjects Over 50 Years of Age
Acronym: SPISAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCAMCFE-00016
Record Dates: First submitted 2020-10-15; First posted 2020-11-02 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2020-10

CONDITIONS: Sarcopenia; Physical Exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group - Spinach (Experimental): Consumption for 90 days of spinach extract (1000mg)
  Four capsules will be consumed per day, two with breakfast and two with lunch.
  Interventions: Dietary Supplement: Dietary supplement consumption and physical exercise
- control group Placebo (sucrose) (Placebo Comparator): Four capsules will be consumed per day, two with breakfast and two with lunch.
  Interventions: Dietary Supplement: Dietary supplement consumption and physical exercise

INTERVENTIONS:
Dietary Supplement: Dietary supplement consumption and physical exercise — The consumption time of the experimental product was 90 days and the control consumption time was 90 days.
  During this time, training should be done three times a week.

SUMMARY:
Controlled, randomized, single-center, double-blind clinical trial, with two parallel branches depending on the product consumed, to measure the efficacy of a supplement extracted from spinach on muscle strength in subjects over 50 years of age.

DETAILED DESCRIPTION:
Subjects who meet the selection criteria will make two visits to the laboratory to perform the tests established in the protocol. In addition, all subjects will develop a program of strength, polyarticular, individualized and progressive exercises in which the main muscle groups are worked. The program will be held three days a week (36 sessions). Subsequently, a statistical analysis will be performed with the variables measured in the study to obtain results.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 75 years.
* Body mass index less than 32.
* Subjects who do not develop physical exercise scheduled on a weekly basis.
* Subjects who have given written informed consent to participate in the study.

Exclusion Criteria:

* Consumption during the 6 months prior to the study of functional food or supplement that modifies body composition.
* Presence of absolute or relative contraindications dictated by the American College of Sports Medicine, for the performance of physical exercise.
* Presence of chronic diseases that prevent the performance of a physical exercise program (disabling arthropathies, moderate / severe chronic lung disease, ischemic heart disease under treatment, arrhythmias, etc.).
* Abuse in the ingestion of alcohol.
* Present hypersensitivity or intolerance to any of the components of the products under study.
* Inability to understand informed consent.
* Serious or terminal illnesses.
* Subjects with a body mass index above 32.
* Pregnant or lactating women.
* Inability to understand informed consent.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Muscle function | From baseline to 90 days
  Isokinetic dynamometry. Knee flexion and extension force
Muscle function | From baseline to 90 days
  Isometric dynamometry

SECONDARY OUTCOMES:
Muscle mass | From baseline to 90 days
  Dual X-ray absorptiometry (DEXA), measured in grams.
Muscle mass | From baseline to 90 days
  Bioimpedance, in grams.
Balance | From baseline to 90 days
  Force platform Kistler
Health Questionnaire | From baseline to 90 days
  Questionnaire Quality of life SF-36. It consists of 36 questions that assess the health and well-being of the person
Nutritional survey | From baseline to 90 days
  24 hour memory
Liver safety variables | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product.
  It is a blood test blood, with the aim of determining if there is any alteration in the liver.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain